CLINICAL TRIAL: NCT07248189
Title: Postoperative Pain After Single Visit Root Canal Treatment Using Commercial or Medical Grade Sodium Hypochlorite as Irrigating Solutions in Patients With Symptomatic Irreversible Pulpitis in Their Mandibular Molars: A Randomized Controlled Trial
Brief Title: The Effect of Commercial and Medical Grade Sodium Hypochlorite on Post Endodontic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maha Nasr, Dr., Egyptian Russian University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ERU3
Record Dates: First submitted 2025-11-18; First posted 2025-11-25 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Symptomatic Irreversible Pulpitis (SIP)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Commercial NaOCl (Active Comparator)
  Interventions: Drug: commercially available Sodium Hypochlorite
- Medical Grade NaOCl (Experimental)
  Interventions: Drug: Medical grade Sodium Hypochlorite

INTERVENTIONS:
Drug: commercially available Sodium Hypochlorite — during the routine root canal treatment of mandibular molars with SIP, irrigation will be performed between each two successive files with 2 ml of half concentration commercially available sodium hypochlorite and after complete preparation 5 ml of the same solution will be used in full concentration for the purpose of smear layer removal.
  Arms: Commercial NaOCl
Drug: Medical grade Sodium Hypochlorite — during the routine root canal treatment of mandibular molars with SIP, irrigation will be performed between each two successive files with 2 ml of half concentration Medical grade sodium hypochlorite and after complete preparation 5 ml of the same solution will be used in full concentration for the purpose of smear layer removal.
  Arms: Medical Grade NaOCl

SUMMARY:
the aim of the current study is to evaluate the effects of commercial and medical formulations of NaOCl on postoperative pain after endodontic treatment of mandibular posterior teeth with acute irreversible pulpitis.

Personal data including name, address, and phone number in addition to medical history and dental history will be collected by the operator from each patient in specific forms, then history of chief complaint will be recorded. The selected patients should show symptoms of irreversible pulpitis. The operator will perform extra-oral and intra-oral clinical examination as the expected tooth to be included in this study should be examined tentatively using a diagnostic mirror and probe. Radiograph will be taken to help to identify if there is widening of periodontal ligament space, periapical radiolucency, deep caries near the pulp chamber or recurrent caries under restoration.

The diagnosis of symptomatic irreversible pulpitis is confirmed through the patients' history of moderate to severe pain with hot and/or cold in mandibular posterior area, prolonged exaggerated response to cold testing than the contralateral tooth and positive response to electric pulp tester. Radiograph should show no or slight widening of periodontal ligaments. After completing the diagnosis (symptomatic irreversible pulpitis) and confirming that the patient fulfills the eligibility criteria, the patient will be enrolled in the study. The treatment will be done in a single visit.

• Treatment procedure: Each patient will be given an NRS chart to rate her /his presenting pain as preoperative pain. After administering anesthesia, access cavity will be performed using round bur size 4 and Endo-Z bur (DENTSPLY, Tulsa Dental, DENTSPLY Maillefer, TN, USA), then the tooth will be isolated using rubber dam, at this point, patients will be randomly assigned to either of two groups according to the used irrigating solution, group 1, irrigation will be done using the professional form of NaOCl and group 2, irrigation will be done using the commercial form of NaOCl. Irrigant preparation will be done by a dentist who is not involved in the study so that the operator would be blind to the irrigant used. Working length will be determined by the apex locator (Root ZX, J.Morita USA, Irvine, USA) and radiographically confirmed as 0.5-1 mm shorter from the radiographic apex. Root canal treatment will be, then, completed using Edge X7 (Edge-Endo, USA) NiTi rotary files system according to the manufacturer instructions. All canals will be thoroughly irrigated using 3ml of 2.5% Sodium hypochlorite between every two subsequent instruments. Canals will be dried then obturated by the modified single cone technique using 0.04 taper gutta percha points and epoxy resin sealer (ADSEAL, METABIOMED.CO., LTD, Korea) and then a spreader will be used to provide space for auxiliary cones. The access cavity will be then sealed with temporary filling (MD-TEMP, META BIOMED CO., LTD. Chungbuuk, Korea).

Patients will be referred to an operative or a fixed prosthodontics specialist for crown placement at the Faculty of Dentistry, Egyptian Russian University. Post-operative instructions and appropriate post-operative rescue medication will be prescribed (400mg Ibuprofen). All patients will be asked to record their postoperative pain level felt on NRS at 6, 12, 24, 48, 72 hours and 7 days.

Research objective (state the aim) The aim of this study is to assess the effect of different sodium hypochlorite preparations (commercial VS medical) on postoperative pain in patients with symptomatic irreversible pulpitis after single visit endodontic treatment.

Sample size:

Anticipated sample size, 60 patients will be included in the study, divided into 2 groups, 30 patients per group.

Grouping & Randomization used:(specify if present) Two groups Group 1: Professional NaOCl Group 2: Commercial NaOCl

Outcome variables:

The primary outcome is the effect on Postoperative pain which will be measured using NRS at 6, 12, 24, 48, 72 hours postoperatively. Numerical Rating Scale (NRS) (20): It is an 11-point scale consisting of numbers from 0 through 10; - 0 reading represents "no pain" - 1-3 readings represent "mild pain" - 4- 6 readings represent "moderate pain" - 7- 10 readings represent "severe pain"

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with symptomatic irreversible pulpitis. 2. Patients with active pain (moderate-to-severe) in mandibular molars. 4. Males and females. 5. Patient with the ability to understand and use pain scales. 6. Patient who accepts to enroll to the study.

Exclusion Criteria:

* 1. Pregnant females. 2. Patients taking pain medication 12 hours earlier. 3. Patient having more than one symptomatic mandibular tooth in the same quadrant.

  4. Patients with periradicular pathosis and/or radiolucency other than widened periodontal ligaments.

  5. Patients with contributory medical history (ASA>II).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-10-01 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-27 (Actual)

PRIMARY OUTCOMES:
Post Operative pain | from enrollemnt to 72 hours after treatment
  incidence and intensity of post operative pain after single visit root canal treatment of mandibular molars with SIP

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Dentistry, Cairo University, Cairo
  - Faculty of Oral and Dental Medicine, Egyptian Russian University, Cairo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Severing AL, Rembe JD, Koester V, Stuermer EK. Safety and efficacy profiles of different commercial sodium hypochlorite/hypochlorous acid solutions (NaClO/HClO): antimicrobial efficacy, cytotoxic impact and physicochemical parameters in vitro. J Antimicrob Chemother. 2019 Feb 1;74(2):365-372. doi: 10.1093/jac/dky432. PMID 30388236
- [Background] van der Waal SV, van Dusseldorp NE, de Soet JJ. An evaluation of the accuracy of labeling of percent sodium hypochlorite on various commercial and professional sources: is sodium hypochlorite from these sources equally suitable for endodontic irrigation? J Endod. 2014 Dec;40(12):2049-52. doi: 10.1016/j.joen.2014.08.021. Epub 2014 Oct 7. PMID 25301349
- [Background] Mostafa MEHAA, El-Shrief YAI, Anous WIO, Hassan MW, Salamah FTA, El Boghdadi RM, El-Bayoumi MAA, Seyam RM, Abd-El-Kader KG, Amin SAW. Postoperative pain following endodontic irrigation using 1.3% versus 5.25% sodium hypochlorite in mandibular molars with necrotic pulps: a randomized double-blind clinical trial. Int Endod J. 2020 Feb;53(2):154-166. doi: 10.1111/iej.13222. Epub 2019 Oct 23. PMID 31563148
- [Background] Siqueira JF Jr, Rocas IN, Favieri A, Machado AG, Gahyva SM, Oliveira JC, Abad EC. Incidence of postoperative pain after intracanal procedures based on an antimicrobial strategy. J Endod. 2002 Jun;28(6):457-60. doi: 10.1097/00004770-200206000-00010. PMID 12067129